CLINICAL TRIAL: NCT04851769
Title: Impact of PCSK9 Inhibitors on Coronary Plaque Composition and Vulnerability in Patients With Coronary Artery Disease Assessed by Optical Coherence Tomography
Brief Title: Impact of PCSK9 Inhibitors on Coronary Plaque Composition and Vulnerability Assessed by Optical Coherence Tomography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Vice president, professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: anzhen201803
Record Dates: First submitted 2021-03-31; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Randomized Controlled Trials
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; alirocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alirocumab plus statin (Experimental): Patients in the alirocumab arm will receive alirocumab 75 mg Q2W added to statin therapy (atorvastatin 20 mg/day or rosuvastatin 10mg/day).
  Interventions: Drug: PCSK9 inhibitor plus statin; Procedure: Coronary imaging follow-up
- standard statin therapy (Active Comparator): Patients in the standard statin arm will continue to receive atorvastatin 20 mg/day or rosuvastatin 10 mg/day. Statin dose escalation or adding concomitant non-statin lipid-lowering therapy could be considered by their responsible physician to achieve an LDL-C target <100 mg/dL.
  Interventions: Drug: standard statin therapy; Procedure: Coronary imaging follow-up

INTERVENTIONS:
Drug: PCSK9 inhibitor plus statin — Patients in the alirocumab arm will receive alirocumab 75 mg Q2W added to statin therapy (atorvastatin 20 mg/day or rosuvastatin 10mg/day).
  Other Names: alirocumab
  Arms: alirocumab plus statin
Drug: standard statin therapy — Patients will continue to receive atorvastatin 20 mg/day or rosuvastatin 10 mg/day.
  Arms: standard statin therapy
Procedure: Coronary imaging follow-up — coronary angiography and OCT imaging at week 36 ± 2 weeks follow-up

SUMMARY:
The study is a prospective, open-label, randomized, single-center study involving patients with intermediate coronary lesions (50%-70% diameter stenosis) and who have elevated LDL-C values (LDL-C≥100 mg/dL) despite stable statin therapy.

Eligible patients are randomized to receive either alirocumab or standard-of-care (1:1). The last dose of alirocumab will be given at week 34. Patients in the alirocumab arm will receive alirocumab 75 mg Q2W added to statin therapy (atorvastatin 20 mg/day or rosuvastatin 10mg/day). Patients in the standard-of-care arm will continue to receive atorvastatin 20 mg/day or rosuvastatin 10 mg/day. OCT images will be acquired at the baseline and at week 36 ± 2 weeks follow-up.

DETAILED DESCRIPTION:
The study is a prospective, open-label, randomized, single-center study involving patients with intermediate coronary lesions (50%-70% diameter stenosis) and who have elevated LDL-C values (LDL-C≥100 mg/dL) despite stable statin therapy.

Eligible patients included those who are (I) at least 18 years of age, (II) diagnosed as stable coronary artery disease or acute coronary syndrome during admission (III) undergoing clinically indicated coronary angiography and identified with at least one intermediate lesion (50%-70% diameter stenosis) on de novo coronary arteries, (IV) have an elevated LDL-C values (LDL-C≥100 mg/dL) despite taken rosuvastatin 10 mg/day or atorvastatin 20 mg/day for 2-4 weeks after initiation or with maximally tolerated statin therapy, (V) able to provide written, informed consent.

The study included a 36-week open-label treatment period (including post-treatment OCT imaging), starting within 4 weeks of baseline coronary angiogram. During the open-label treatment period, patients are randomized to receive either alirocumab or standard-of-care (1:1). The last dose of alirocumab will be given at week 34.

Patients in the alirocumab arm will receive alirocumab 75 mg Q2W added to statin therapy (atorvastatin 20 mg/day or rosuvastatin 10mg/day). Patients in the standard-of-care arm will continue to receive atorvastatin 20 mg/day or rosuvastatin 10 mg/day. Statin dose escalation or adding concomitant non-statin lipid-lowering therapy would be considered by their responsible physician to achieve an LDL-C target <100 mg/dL. Antithrombotic therapy and other concomitant medications are exclusively decided by the responsible physicians. Follow-up coronary angiograms and OCT imaging analyses of the same vessels will be carried out at the end of treatment period (at week 36 ± 2 weeks, depending on patient availability) in both study arms. Regular medical examination and laboratory tests will be conducted at weeks 4, 12, 24, and 36. All enrolled patients are monitored and evaluated for safety and any other adverse events during the study period.

ELIGIBILITY:
Inclusion Criteria:

(I) 18 - 80 years of age, (II) diagnosed as stable coronary artery disease or acute coronary syndrome during admission (III) undergoing clinically indicated coronary angiography and identified with at least one intermediate lesion (50%-70% diameter stenosis) on de novo coronary arteries, (IV) have an elevated LDL-C values (LDL-C≥100 mg/dL) despite taken rosuvastatin 10 mg/day or atorvastatin 20 mg/day for 2-4 weeks after initiation or with maximally tolerated statin therapy, (V) able to provide written, informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with at least one dose of any anti-PCSK9 monoclonal antibody
2. received target vessel revascularization
3. Known hypersensitivity or have contraindications to any anti-PCSK9 monoclonal antibody or statins
4. Unable to receive OCT imaging tests
5. Known history of hemorrhagic stroke
6. Currently under treatment for cancer
7. Baseline triglyceride > 400 mg/dl
8. Patients with severe liver or renal dysfunction
9. Pregnant or breast-feeding women
10. Considered by the investigator as inappropriate for this study for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
minimum fibrous-cap thickness | 36 weeks
  The primary endpoint of the study is the OCT derived changes in minimum fibrous-cap thickness between baseline and follow-up.

SECONDARY OUTCOMES:
minimum lumen area and maximum lipid arc | 36 weeks
  Secondary endpoints include minimum lumen area between baseline and follow-up, as well as the absolute changes in maximum lipid arc.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao F, Li YP, Ma XT, Wang ZJ, Shi DM, Zhou YJ. Effect of Alirocumab on Coronary Calcification in Patients With Coronary Artery Disease. Front Cardiovasc Med. 2022 May 6;9:907662. doi: 10.3389/fcvm.2022.907662. eCollection 2022. PMID 35600486
- [Derived] Gao F, Wang ZJ, Ma XT, Shen H, Yang LX, Zhou YJ. Effect of alirocumab on coronary plaque in patients with coronary artery disease assessed by optical coherence tomography. Lipids Health Dis. 2021 Sep 12;20(1):106. doi: 10.1186/s12944-021-01528-3. PMID 34511134